CLINICAL TRIAL: NCT00001851
Title: Evaluation and Treatment to Improve Bone Quality and Prevent Fractures by the Percutaneous Replacement of Diseased Tissue in Polyostotic Fibrous Dysplasia and McCune-Albright Syndrome
Brief Title: Bone Marrow Injection to Replace Diseased Bone in Polyostotic Fibrous Dysplasia and McCune-Albright Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990003; 99-D-0003
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-06-26

CONDITIONS: Polyostotic Fibrous Dysplasia
Keywords: Marrow; Grafting; Imaging; Injection; Aspiration; Bone Marrow Stromal Cells; Bone Grafting; Bone Graft Substitutes; Bio and Pharmacological Regulators of Bone Turnover
MeSH Terms: conditions — Fibrous Dysplasia, Polyostotic

SUMMARY:
This study will evaluate the effectiveness of a new bone injection technique for treating bone disease in patients with polyostotic fibrous dysplasia or McCune-Albright syndrome. In these patients, some bones develop areas with much less mineral, making the bones more prone to fracture or deformity and causing pain. This new treatment is intended to reduce the risk of fracture, minimize deformities and improve overall function in these patients.

Patients 4 years of age and older with bone lesions that are highly likely to cause significant pain and illness may be eligible for this 2-year study. Participants must be simultaneously enrolled in NIDCR's research protocol 98-D-0145 (Screening and Natural History of Patients with Polyostotic Fibrous Dysplasia and McCune-Albright Syndrome) or 98-D-0146 (A Randomized, Placebo-Controlled Trial of Alendronate in the Treatment of Polyostotic Fibrous Dysplasia and McCune-Albright Syndrome).

Within 14 days of the bone injection procedure, patients will have a medical history, routine blood tests, urinalysis and check of vital signs (blood pressure, pulse and temperature) and will complete a 30-minute quality-of-life questionnaire. Women of child-bearing potential will have a pregnancy test. Patients who do not have recent X-rays and bone density scans available for review will have new ones taken. When these studies are completed, patients will undergo the bone injection procedure, followed immediately by bone densitometry and coned-down X-rays, as follows:

* Bone injection - Patients will be given an anesthetic either to make them sleepy or put them to sleep completely. A portion of bone marrow will be withdrawn through a needle inserted into the hip bone and, at the same time, abnormal bone in the arms and legs will be sucked out using a needle. The abnormal bone will be replaced with a mixture of bone marrow and collagen (connective tissue protein) injected into the hole in the bone. The areas of injection will be closed
* Bone densitometry - X-rays of the operated bone and opposite normal bone will be taken.
* Coned-down X-rays - Magnified normal X-rays will be taken as close-ups of an active lesion.

Patients will have a history and physical examination by their local physician or at NIH every month for the first 4 months after the procedure. Every 6 months after the procedure, patients will return to NIH for follow-up, including a physical examination and completion of a quality-of-life questionnaire. Imaging studies of the injected site will be done 3, 6, and 12 months after the procedure.

DETAILED DESCRIPTION:
Polyostotic fibrous dysplasia (PFD) is a sporadic disorder which affects multiple sites in the skeleton. The bone at these sites is rapidly resorbed and replaced by abnormal fibrous tissue. PFD may occur alone or as part of the McCune-Albright Syndrome (MAS), a syndrome originally defined by the triad of PFD, cafe au lait pigmentation of the skin, and precocious puberty. The bony lesions are frequently disfiguring and painful. In addition, depending on the location of the lesion, they can cause significant morbidity. Lesions in weight-bearing bones can lead to disabling fractures, while lesions in the skull can lead to compression of vital structures such as the cranial nerves.

Currently there are no clearly-defined systemic or local therapies for the bone disease, and results of the use of conventional surgical treatment of sites of impending fracture have been universally disappointing. In this study, we will treat osteolytic lesions in the long bones of the upper and lower extremities, the sites of potential fracture, with a novel surgical approach. This will involve 1) the removal of abnormal tissue through percutaneous aspiration, and 2) the use of skeletal precursor cells taken from the unaffected sites, mixed with a bone grafting substitute, and injected into the affected sites to bring about an improvement in local bone quality and overall patient function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be otherwise healthy women, men, and children, with polyostotic fibrous dysplasia (PFD)/McCune-Albright Syndrome (MAS).

Children will be greater than 4 years of age.

The diagnosis will be based on evidence of the clinical spectrum of the disease and confirmed by the presence of typical findings on bone biopsy.

All patients must be actively enrolled in the Screening and Natural History Protocol and possibly the Bisphosphonate Protocol.

Patients will be enrolled in the study if they have a lytic lesion of the humerus, femur, or tibia which satisfies at least one of the following criteria: the lesion encompasses at least 50% of the width of the bone at that point on both AP and lateral radiographs; the lesion has caused a change in the anatomical shape and contour of the bone; the lesion has a bone density less than 50% of the density of the contralateral, normal side.

Patients on previous or concomitant therapy are eligible for enrollment.

Patients on the Bisphosphonate Protocol must have received at least one month of treatment on that protocol before receiving a bone marrow injection in this protocol.

Women in childbearing age will be offered barrier methods of contraception to decrease the risk of pregnancy for a period of one year following the transplant. Subjects who become pregnant during year one of the study will be transferred to the inactive participant group. Pregnancy testing will be performed prior to research procedures and surgery. Subjects using oral contraceptive agents are included. Women without normal menstrual cycles will be offered hormone replacement therapy for a period of 3 cycles prior to treatment.

Subjects must agree to travel to NIH during the first 24 months and remain in the Bethesda area for the post-operative period as defined by protocol requirements.

EXCLUSION CRITERIA:

Subjects will be excluded if they receive phenobarbital or related antiepileptic agents, including Dilantin or Tegretol.

Medical problems which will preclude participation in the study include: pregnancy; chronic or active dermatological disease; chronic anemia (thalassemia, etc.); diabetes mellitus (fasting blood glucose in excess of 140 mg/dl); active or chronic pulmonary disease including COPD, chronic bronchitis, or asthma requiring medications; active or chronic gastrointestinal disease including gastric and duodenal ulcer disease and inflammatory bowel disease; history of cancer except for dermal lesions; intestinal malabsorption, chronic or active renal disease including a serum creatinine above 1.8 mg/dl; chronic or active hepatic disease including hepatitis; HIV infection.

Subjects may not smoke more than one pack of cigarettes per day.

Alcohol consumption must be less than 1.5 oz per day, without binge drinking.

Subjects should have no dietary aberrations and no history of anorexia nervosa within the past 10 years.

Subjects must be willing to receive transfusions of blood products if it is deemed medically necessary to preserve their well-being or their life.

Patients will be excluded if they have a history of an allergy to all of the following antibiotics: penicillin, tetracycline, and cephalosporins.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1998-12-15; Primary Completion 2002-04-30 (Actual); Study Completion 2002-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Danon M, Crawford JD. The McCune-Albright syndrome. Ergeb Inn Med Kinderheilkd. 1987;55:81-115. doi: 10.1007/978-3-642-71052-0_3. No abstract available. PMID 3545811
- [Background] Mastorakos G, Mitsiades NS, Doufas AG, Koutras DA. Hyperthyroidism in McCune-Albright syndrome with a review of thyroid abnormalities sixty years after the first report. Thyroid. 1997 Jun;7(3):433-9. doi: 10.1089/thy.1997.7.433. PMID 9226216
- [Background] Mauras N, Blizzard RM. The McCune-Albright syndrome. Acta Endocrinol Suppl (Copenh). 1986;279:207-17. doi: 10.1530/acta.0.112s207. PMID 3465162